CLINICAL TRIAL: NCT03192189
Title: Development of a Decision-making Aid for Referring Severe Kidney Injury Patients for Nephrology Consultations
Acronym: IRA Cible
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2016/OM-01
Record Dates: First submitted 2017-06-16; First posted 2017-06-20 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Diseases; Acute Kidney Injury
MeSH Terms: conditions — Renal Insufficiency, Chronic; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute kidney injury: Requiring treatment with dialysis
  Interventions: Other: monitoring for progression to chronic kidney disease

INTERVENTIONS:
Other: monitoring for progression to chronic kidney disease — Collect clinical information and assess risk factors

SUMMARY:
Acute kidney injury is a frequent and growing complication associated with a risk of progressing into a chronic kidney disease. Recent guidelines have recommended systematic consultations with a nephrologist 3-6 months following hospitalization. Risk factors of developing chronic kidney disease between hospital visits are understudied.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Suffering from acute kidney injury treated with dialysis
* hospitalized in a university center from August 2016 to December 2017 with severe AKI defined according to 2 of the 3 criterion definitions of KDIGO stage AKI: an increase in SCr above 354 μmol/Lor renal replacement therapy (RRT) indication, but not the 3-fold increase in SCr increase within 7 days with SCr below 354 μmol/L.
* The patient has been informed and does not oppose the study
* The patient is insured or the beneficiary of a health insurance policy

Exclusion Criteria:

* The patients is under judicial protection or state guardianship
* Patient has chronic kidney disease(CKD) KDIGO stage 5
* It proves impossible to give the patient clear information
* patients living with kidney transplant
* plan dialysis for bilateral surgery nephrectomy
* patient refuse to participate and patients with no health insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing dialysis for acute kidney injury. All new adults (>18 years old) hospitalized in a university center with severe AKI was included from August 2016 to December 2017. Inclusion criteria was a severe AKI defined by dialysis start for AKI or an increase of Scr upper 354 μmol/L. Exclusion criteria was CKD stage 5 , patients living with kidney transplant, plan dialysis for bilateral surgery nephrectomy, patient witch justice protection and refuse to participate. Eligible patients were identified by physicians for ICU and nephrology department and by laboratory biochemistry department for others wards. A Biochemistry alert system controlled the exhaustively of inclusion in ICU and Nephrology department during the period of the study.
Sampling Method: Non-Probability Sample
Enrollment: 319 (Actual)
Dates: Start 2016-08-20 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Develop a prognostic score of progression to chronic kidney disease at 6 months in patients requiring hospitalization for dialysis for acute kidney injury to identify those who would benefit from consultation with a nephrologist | 6 months

SECONDARY OUTCOMES:
Identify new risk factors for progression to chronic kidney disease at 6 months post dialysis for acute kidney injury pre-hospitalization and during hospitalization and day of discharge | 6 months
Identify renal phenotype of patients with chronic kidney disease | 6 months
  characterization from renal biopsy
Evaluate mortality during hospital stay | 1 months
Evaluate mortality at medium-term | 6 months
Identify specific therapeutic interventions put into place during the 6 month consultation | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cardinale A, Messikh Z, Antoine V, Aglae C, Reboul P, Cariou S, Muller L, Lefrant JY, Moranne O. Specificity of severe AKI aetiology and care in the elderly. The IRACIBLE prospective cohort study. J Nephrol. 2022 Nov;35(8):2097-2108. doi: 10.1007/s40620-022-01322-z. Epub 2022 May 3. PMID 35503200